CLINICAL TRIAL: NCT01676909
Title: A Hybrid Effectiveness-Implementation Trial of a Wellness Self-Management Program
Brief Title: Wellness Self-Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 11-276
Record Dates: First submitted 2012-07-02; First posted 2012-08-31 (Estimated); Results first posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-02

CONDITIONS: Mental Illness; Chronic Medical Illness
Keywords: self-management
MeSH Terms: conditions — Mental Disorders | interventions — Self-Help Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Living Well (Experimental): This study will involve a clinical trial of Living Well (LW), a 12-session, peer co-led, group intervention designed to help veterans with co-occurring Serious Mental Illnesses and Chronic Medical Conditions learn techniques for better health management and ways to live a healthier lifestyle. Key topics that will be discussed are medication side effects, how symptoms of mental illness may affect veterans' ability to manage their medical conditions, effects of substance use on medical and mental health functioning, learning ways to eat healthier and exercise, and how to communicate more effectively with care providers. After completing the 12 weekly groups, participants will return to complete once monthly booster group sessions for the next three months.
  Interventions: Behavioral: Living Well
- Medical Illness Education & Support Group (Active Comparator): We selected a comparison condition that would provide parallel focus (i.e. medical illness) but not include use of the core ingredients undergirding the Living Well intervention including behavioral action planning, problem solving, in-session and between session practice using specific disease self-management techniques and involvement of peer co-facilitators to enhance modeling and improve self-efficacy and activation. As with Living Well, the content of the intervention will have broad applicability across diverse chronic disease conditions. The comparison condition will be a once-weekly support and education group focusing on living with a chronic medical condition.
  Interventions: Behavioral: Medical Illness Education & Support Group

INTERVENTIONS:
Behavioral: Living Well — This study will involve a clinical trial of Living Well (LW), a 12-session, peer co-led, group intervention designed to help veterans with co-occurring Serious Mental Illnesses and Chronic Medical Conditions learn techniques for better health management and ways to live a healthier lifestyle. Key topics that will be discussed are medication side effects, how symptoms of mental illness may affect veterans' ability to manage their medical conditions, effects of substance use on medical and mental health functioning, learning ways to eat healthier and exercise, and how to communicate more effectively with care providers. There will be 3 booster sessions after the 12 sessions, once a month for 3 months.
  Arms: Living Well
Behavioral: Medical Illness Education & Support Group — The comparison condition will be a general Medical Illness Education and Support (MIES) group that will discuss common challenges experienced by those living with a wide range of chronic illnesses and behavioral and lifestyle management techniques that may help veterans to better handle chronic medical conditions that also meets for 12 weeks.
  Arms: Medical Illness Education & Support Group

SUMMARY:
Veterans with schizophrenia, other serious mental illnesses (SMI), and Post Traumatic Stress Disorder (PTSD) are at elevated risk for co-occurring chronic medical conditions resulting in increased risk of disability, high health care spending, reduced quality of life and early mortality. Physical wellness is increasingly recognized as a key component of the VA's commitment to developing recovery-oriented and Veteran-centered mental health treatment. There is also growing recognition of the value of interventions that promote and improve patient self-management of chronic medical conditions. Building on the established efficacy of consumer facilitated medical illness self-management programming used in the general population and two recent adaptations for use with SMI adults in the public health sector (including the investigators' own evaluation of an intervention called Living Well), the investigators propose to complete a randomized controlled effectiveness trial of the Living Well intervention and simultaneously conduct a well specified process evaluation to optimize knowledge accrual regarding important factors that may improve future adoption, implementation and sustainability of the Living Well intervention in the VA system of care.

DETAILED DESCRIPTION:
Background:

Veterans with schizophrenia, other serious mental illnesses (SMI), and Post Traumatic Stress Disorder (PTSD) are at elevated risk for co-occurring chronic medical conditions resulting in increased risk of disability, high health care spending, reduced quality of life and early mortality. Physical wellness is increasingly recognized as a key component of the VA's commitment to developing recovery-oriented and Veteran-centered mental health treatment. There is also growing recognition of the value of interventions that promote and improve patient self-management of chronic medical conditions. Building on the established efficacy of consumer facilitated medical illness self-management programming used in the general population and two recent adaptations for use with SMI adults in the public health sector (including the investigators' own evaluation of an intervention called Living Well), the investigators propose to complete a randomized controlled effectiveness trial of the Living Well intervention and simultaneously conduct a well specified process evaluation to optimize knowledge accrual regarding important factors that may improve future adoption, implementation and sustainability of the Living Well intervention in the VA system of care.

Aims:

Primary AIM 1: Complete a randomized controlled effectiveness trial of the Living Well intervention with 242 Veterans with mental illness and at least one co-occurring chronic medical condition and evaluate the intervention's effects on functional and service related outcomes. The investigators hypothesize that those randomized to the Living Well intervention will, in comparison to those randomized to a medical illness education and support group, demonstrate improved general health functioning including physical and emotional functioning as well as reduced rates of medical emergency room visits for management of a chronic medical condition. The investigators will also evaluate intervention effects on more proximal attitudinal and behavioral outcomes and assess how these factors mediate improvement in the functional and services related outcomes.

Primary AIM 2: Complete a well specified process evaluation based on the RE-AIM evaluation framework to better understand contextual factors that can improve the Reach, Effectiveness, Adoption, Implementation and Maintenance which together determine the potential public health impact of the Living Well intervention.

Methods:

A mix of temporally overlapping quantitative and qualitative methods will be used to maximize integration and synthesis of data streams across the two aims to optimize knowledge accrual.

Impact:

Despite the growing recognition that self-management strategies hold enormous promise for improving quality and outcomes of care for chronic medical illnesses, and the fact that self-management is gaining prominence as a mental health recovery oriented treatment focus, there are currently no evidence-based peer facilitated medical illness self-management interventions available for dissemination within the VA mental health system. The proposed study is designed to both generate evidence supporting the effectiveness of a peer co-facilitated intervention and to help speed throughput to public health impact by collecting important contextual information about factors that may improve future dissemination and implementation efforts.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of schizophrenia/ schizoaffective disorder
* bipolar disorder
* major depression with psychotic features
* post traumatic stress disorder
* or psychosis not otherwise specified (NOS)
* age between 18 and 80
* chart documented presence of at least one of the following chronic medical conditions:

  * a respiratory condition (e.g. asthma, COPD)
  * diabetes
  * arthritis
  * cardiovascular condition (e.g. congestive heart failure, hypertension, etc.)
* receiving mental health services at a designated study site
* willing and able to provide consent to participate
* deemed clinically stable enough to participate in the study by a treatment provider

Exclusion Criteria:

* Severe or profound mental retardation
* Because participants must be able to attend the intervention if assigned to either condition, we will also require potential participants to verify their availability during screening
* Participation in current ongoing study 'Reducing Internalized Stigma in People with Serious Mental Illness"

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Goldberg, PhD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (2):
- United States (2):
  - Washington DC VA Medical Center, Washington, DC, Washington D.C., District of Columbia
  - Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Muralidharan A, Peeples A, Lucksted A. Health Behavior Change Processes Among Adults With Serious Mental Illness Engaged in Illness Self-Management. Qual Health Res. 2021 May;31(6):1155-1168. doi: 10.1177/1049732321992049. Epub 2021 Feb 15. PMID 33588639

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 262 participants were enrolled in the study prior to randomization. 20 participants were not able to be randomized due to attrition resulting in a final study sample of 242.
Groups:
- Living Well: Living Well (LW) will be implemented as a 12-session, peer co-led, group intervention (4-8 persons) designed to help veterans with co-occurring Serious Mental Illnesses and Chronic Medical Conditions learn techniques for better health management and ways to live a healthier lifestyle. Key topics that will be discussed are medication side effects, how symptoms of mental illness may affect veterans' ability to manage their medical conditions, effects of substance use on medical and mental health functioning, learning ways to eat healthier and exercise, and how to communicate more effectively with care providers. Groups will meet weekly for 75 minutes for three months (12 sessions). There will be 3 booster sessions after the 12 sessions, once a month for 3 months.
- Medical Illness Education and Support Group: The comparison condition, Medical Illness Education and Support (MIES) group, will discuss common challenges experienced by those living with a wide range of chronic illnesses and behavioral and lifestyle management techniques that may help veterans to better handle chronic medical conditions. Each of the 12 sessions will follow a basic structure that includes a review of the material presented in the previous session, new education content and discussion.
Period: Overall Study
Arm/Group | Living Well | Medical Illness Education and Support Group
Started | 124 | 118
Post-Treatment Assessment | 105 (19 not completed (3 withdrawn, 15 timed out, 1 declined)) | 107 (11 not completed (5 withdrawn, 6 timed out))
Completed | 106 (18 not completed (3 withdrawn, 15 timed out)) | 104 (14 not completed (5 withdrawn, 9 timed out)
Not Completed | 18 | 14
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Lost to Follow-up | 15 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Living Well | Medical Illness Education and Support Group | Total
Number analyzed (Participants) | 124 | 118 | 242
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (7.6) | 57.0 (7.8) | 57.8 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 32
  Male | 107 | 103 | 210
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 118 | 117 | 235
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 82 | 69 | 151
  White | 31 | 38 | 69
  More than one race | 11 | 11 | 22
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Short Form-12 (SF-12) General Health (Norm Based)
Description: 12-item Short-Form Health Survey. Possible subscale scores range from 0 to 100, with higher scores indicating greater well-being.The SF-12 (39), a widely used standardized instrument with strong psychometric properties, will be used to assess self-perceptions of general health functioning across multiple dimensions (including general, physical and emotional/psychiatric functioning). The SF-12 has shown good internal, consistency, stability, and concurrent validity in outpatients with serious mental illness.
Time Frame: Baseline, Post-intervention (3 months after baseline)
Population: Due to participant attrition, the number of participants analyzed at each time point decreased from the original baseline number.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Living Well | Medical Illness Education and Support Group
Number analyzed (Participants) | 124 | 118
units on a scale
  Baseline | 40.4 (12.0) | 38.9 (12.5)
  Post-intervention: number analyzed (Participants) | 105 | 107
  Post-intervention | 42.5 (11.3) | 41.6 (12.2)
Statistical Analysis 1: Comparison: Living Well vs Medical Illness Education and Support Group; To test hypothesis 1, regarding the three SF-12 subscales, a linear mixed effects models was used. All available data were used from all three assessment time points. Group, time, and group-by-time terms were included in the model. To test for a group difference in mean change from baseline to post-intervention, the significance test of the group-by-post-intervention coefficient was performed. A logistic mixed model for change in proportion with an ED visit was used to test hypothesis 2; Test type: Superiority; p = 0.362, Mixed Models Analysis

2. Primary Outcome: Short-Form 12 (SF-12) Physical Scale (Norm Based)
Description: 12-item Short-Form Health Survey. Possible subscale scores range from 0 to 100, with higher scores indicating greater well-being. The SF-12 , a widely used standardized instrument with strong psychometric properties, will be used to assess self-perceptions of general health functioning across multiple dimensions (including general, physical and emotional/psychiatric functioning). The SF-12 has shown good internal, consistency, stability, and concurrent validity in outpatients with serious mental illness.
Time Frame: Baseline, Post-intervention (3 months after baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Living Well | Medical Illness Education and Support Group
Number analyzed (Participants) | 124 | 118
units on a scale
  Baseline | 39.2 (10.4) | 38.6 (11.4)
  Post-intervention: number analyzed (Participants) | 105 | 107
  Post-intervention | 39.0 (10.3) | 40.2 (11.3)
Statistical Analysis 1: Comparison: Living Well vs Medical Illness Education and Support Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.026, Mixed Models Analysis

3. Primary Outcome: Short-Form 12 (SF-12) Mental Scale (Norm Based)
Description: as for outcome 2
Time Frame: Baseline, Post-intervention (3 months after baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Living Well | Medical Illness Education and Support Group
Number analyzed (Participants) | 124 | 118
units on a scale
  Baseline | 41.3 (11.9) | 40.7 (11.5)
  Post-intervention: number analyzed (Participants) | 105 | 107
  Post-intervention | 44.0 (11.4) | 40.5 (11.6)
Statistical Analysis 1: Comparison: Living Well vs Medical Illness Education and Support Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.032, Mixed Models Analysis

4. Primary Outcome: ER Visit Between Baseline and the 6-month Follow-up
Description: Emergency Room Visit during the approximate 6-month period between baseline and the follow-up visit.
Time Frame: Baseline, Follow-up (6-months after baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | Living Well | Medical Illness Education and Support Group
Number analyzed (Participants) | 124 | 118
Participants
  Baseline | 49 | 45
  6 month follow-up | 47 | 48
Statistical Analysis 1: Comparison: Living Well vs Medical Illness Education and Support Group; A logistic mixed effects model over two 6-month time periods (prior to baseline and between baseline and the 6-month follow-up visit) was used. Terms in the model included group, binary time (pre-f/u versus pre-baseline), and group by time interaction. Two-sided alpha = .05 level tests were used. The hypothesis that the proportion with ER visits would decrease in the Living Well group versus the control group was tests by test of the interaction term; Test type: Superiority; p = .64, Mixed Models Analysis

5. Secondary Outcome: Illness Management Self-Efficacy
Description: This questionnaire is based on the items used in the original Chronic Disease Self-Management Program (CDSMP) as part of that groups extensive evaluation of the curriculum. The original CDSMP measure has been shown to have strong test-retest reliability and internal consistency as well. This subscale consists of 2 items with possible responses ranging from Never (0) to Always (5). Combined scores from these 2 items may range from 0-10 on this subscale, higher scores indicating greater frequency.
Time Frame: Baseline, Post-intervention (3 months after baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Living Well | Medical Illness Education and Support Group
Number analyzed (Participants) | 124 | 118
units on a scale
  Baseline | 5.5 (2.1) | 5.5 (2.0)
  Post-intervention: number analyzed (Participants) | 105 | 107
  Post-intervention | 6.2 (1.9) | 5.4 (2.1)
Statistical Analysis 1: Comparison: Living Well vs Medical Illness Education and Support Group; The same mixed model used for testing hypothesis 1 was used to test treatment effects on secondary scale outcomes (Hypothesis 3: health-related self-efficacy, patient activation; Hypothesis 4: six subscales of the Measure of Self-Management Behaviors) and several other pre-specified outcomes. To test for a group difference in mean change from baseline to follow-up (hypothesis 5) on all primary and secondary outcomes, the significance test of the group-by-follow-up coefficient was performed; Test type: Superiority; p < .0001, Mixed Models Analysis

6. Secondary Outcome: Patient Activation Measure
Description: This 13-item questionnaire measures an individual's perceived ability to manage his or her illness and health behaviors and act as an effective patient. Responses range from Disagree Strongly (1) to Agree Strongly (4). Respondents must complete at least 10 of the 13 questions to obtain a reliable score. Scores may range from 0-100 with higher scores interpreted as greater ability to manage one's own illness. The measure has demonstrated reliability and validity.
Time Frame: Baseline, Post-intervention (3 months after baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Living Well | Medical Illness Education and Support Group
Number analyzed (Participants) | 124 | 118
units on a scale
  Baseline | 60.8 (15.2) | 58.8 (14.6)
  Post-intervention: number analyzed (Participants) | 105 | 107
  Post-intervention | 64.3 (14.0) | 58.9 (14.3)
Statistical Analysis 1: Comparison: Living Well vs Medical Illness Education and Support Group; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.038, Mixed Models Analysis

7. Secondary Outcome: Measure of Self-Management Behaviors - General Self-Management Behaviors Subscale
Description: This questionnaire is based on the items used in the original CDSMP as part of that groups extensive evaluation of the curriculum. The original CDSMP measure has been shown to have adequate psychometric properties; the range of test-retest coefficients for the original illness management scales was .56 to .92, with internal-consistency coefficients ranging from .70 to .75. The General Self-Management Behaviors Subscale consists of 2 items with responses ranging from Never (0) to Always (5). Combined scores from these 2 items may range from 0-10 on this subscale, higher scores indicating greater frequency of using the behavior indicating greater self-management behavior.
Time Frame: Baseline, Post-intervention (3 months after baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Living Well | Medical Illness Education and Support Group
Number analyzed (Participants) | 124 | 118
units on a scale
  Baseline | 2.7 (1.1) | 2.3 (1.2)
  Post-intervention: number analyzed (Participants) | 105 | 107
  Post-intervention | 2.9 (1.2) | 2.6 (1.2)
Statistical Analysis 1: Comparison: Living Well vs Medical Illness Education and Support Group; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.544, Mixed Models Analysis

8. Secondary Outcome: Measure of Self-Management Behaviors - Making Better Use of Health Care Subscale
Description: This questionnaire is based on the items used in the original CDSMP as part of that groups extensive evaluation of the curriculum. The original CDSMP measure has been shown to have adequate psychometric properties; the range of test-retest coefficients for the original illness management scales was .56 to .92, with internal-consistency coefficients ranging from .70 to .75. The Making Better Use of Health Care Subscale consists of 4 items with responses ranging from Never (0) to Always (5).Combined scores from these 4 items may range from 0-20 on this subscale, higher scores indicating greater frequency of using the behavior indicating greater self-management behavior.
Time Frame: Baseline, Post-intervention (3 months after baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Living Well | Medical Illness Education and Support Group
Number analyzed (Participants) | 124 | 118
units on a scale
  Baseline | 2.9 (1.4) | 2.5 (1.4)
  Post-intervention: number analyzed (Participants) | 105 | 107
  Post-intervention | 3.3 (1.2) | 2.9 (1.3)
Statistical Analysis 1: Comparison: Living Well vs Medical Illness Education and Support Group; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.699, Mixed Models Analysis

9. Secondary Outcome: Measure of Self-Management Behaviors - Behavioral and Cognitive Symptom Management Subscale
Description: This questionnaire is based on the items used in the original CDSMP as part of that groups extensive evaluation of the curriculum. The original CDSMP measure has been shown to have adequate psychometric properties; the range of test-retest coefficients for the original illness management scales was .56 to .92, with internal-consistency coefficients ranging from .70 to .75. The Behavioral and Cognitive Symptom Management Subscale consists of 6 items with responses ranging from Never (0) to Always (5). Combined scores from these 4 items may range from 0-30 on this subscale, higher scores indicating greater frequency or using the behavior indicating greater self-management.
Time Frame: Baseline, Post-intervention (3 months after baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Living Well | Medical Illness Education and Support Group
Number analyzed (Participants) | 124 | 118
units on a scale
  Baseline | 2.2 (1.1) | 2.2 (1.0)
  Post-intervention: number analyzed (Participants) | 105 | 107
  Post-intervention | 2.5 (1.0) | 2.2 (0.9)
Statistical Analysis 1: Comparison: Living Well vs Medical Illness Education and Support Group; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.006, Mixed Models Analysis

10. Secondary Outcome: Measure of Self-Management Behaviors - Accessing Social Support Subscale
Description: This questionnaire is based on the items used in the original CDSMP as part of that groups extensive evaluation of the curriculum. The original CDSMP measure has been shown to have adequate psychometric properties; the range of test-retest coefficients for the original illness management scales was .56 to .92, with internal-consistency coefficients ranging from .70 to .75. The Accessing Social Support Subscale consists of 2 items with responses ranging from Never (0) to Always (5). Combined scores from these 2 items may range from 0-10 on this subscale, higher scores indicating greater frequency of using the behavior indicating greater self-management behavior.
Time Frame: Baseline, Post-intervention (3 months after baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Living Well | Medical Illness Education and Support Group
Number analyzed (Participants) | 124 | 118
units on a scale
  Baseline | 2.3 (1.4) | 2.3 (1.2)
  Post-intervention: number analyzed (Participants) | 105 | 107
  Post-intervention | 2.4 (1.3) | 2.4 (1.3)
Statistical Analysis 1: Comparison: Living Well vs Medical Illness Education and Support Group; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.762, Mixed Models Analysis

11. Secondary Outcome: Measure of Self-Management Behaviors - Physical Activity Subscale
Description: This questionnaire is based on the items used in the original CDSMP as part of that groups extensive evaluation of the curriculum. The original CDSMP measure has been shown to have adequate psychometric properties; the range of test-retest coefficients for the original illness management scales was .56 to .92, with internal-consistency coefficients ranging from .70 to .75. The Physical Activity Subscale consists of 2 items with responses ranging from Never (0) to Always (5). Combined scores from these 2 items may range from 0-10 on this subscale, higher scores indicating greater frequency of using the behavior indicating greater self-management behavior.
Time Frame: Baseline, Post-intervention (3 months after baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Living Well | Medical Illness Education and Support Group
Number analyzed (Participants) | 124 | 118
units on a scale
  Baseline | 2.3 (1.3) | 2.3 (1.3)
  Post-intervention: number analyzed (Participants) | 105 | 107
  Post-intervention | 2.7 (1.3) | 2.4 (1.3)
Statistical Analysis 1: Comparison: Living Well vs Medical Illness Education and Support Group; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.326, Mixed Models Analysis

12. Secondary Outcome: Measure of Self-Management Behaviors - Healthy Eating Subscale
Description: This questionnaire is based on the items used in the original CDSMP as part of that groups extensive evaluation of the curriculum. The original CDSMP measure has been shown to have adequate psychometric properties; the range of test-retest coefficients for the original illness management scales was .56 to .92, with internal-consistency coefficients ranging from .70 to .75. The Healthy Eating Subscale consists of 2 items with responses ranging from Never (0) to Always (5). Combined scores from these 2 items may range from 0-10 on this subscale, higher scores indicating greater frequency of using the behavior indicating greater self-management behavior.
Time Frame: Baseline, Post-intervention (3 months after baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Living Well | Medical Illness Education and Support Group
Number analyzed (Participants) | 124 | 118
units on a scale
  Baseline | 2.6 (1.3) | 2.5 (1.3)
  Post-intervention: number analyzed (Participants) | 105 | 107
  Post-intervention | 3.0 (1.1) | 2.7 (1.1)
Statistical Analysis 1: Comparison: Living Well vs Medical Illness Education and Support Group; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.667, Mixed Models Analysis

13. Secondary Outcome: Short Form-12 (SF-12) General Health (Norm Based)
Description: as for outcome 1
Time Frame: Baseline, Post-Intervention (3 months after baseline), Follow-Up (6 months after baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Living Well | Medical Illness Education and Support Group
Number analyzed (Participants) | 124 | 118
units on a scale
  Baseline | 40.4 (12.0) | 38.9 (12.5)
  Post-intervention: number analyzed (Participants) | 105 | 107
  Post-intervention | 42.5 (11.3) | 41.6 (12.2)
  Follow-up: number analyzed (Participants) | 106 | 104
  Follow-up | 42.9 (12.0) | 39.2 (12.2)
Statistical Analysis 1: Comparison: Living Well vs Medical Illness Education and Support Group; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.142, Mixed Models Analysis

14. Secondary Outcome: Short-Form 12 (SF-12) Physical Scale (Norm Based)
Description: as for outcome 2
Time Frame: Baseline, Post-Intervention (3 months after baseline), Follow-Up (6 months after baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Living Well | Medical Illness Education and Support Group
Number analyzed (Participants) | 124 | 118
units on a scale
  Baseline | 39.2 (10.4) | 38.6 (11.4)
  Post-intervention: number analyzed (Participants) | 105 | 107
  Post-intervention | 39.0 (10.3) | 40.2 (11.3)
  Follow-up: number analyzed (Participants) | 106 | 104
  Follow-up | 40.3 (10.2) | 38.4 (12.3)
Statistical Analysis 1: Comparison: Living Well vs Medical Illness Education and Support Group; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.342, Mixed Models Analysis

15. Secondary Outcome: Short-Form 12 (SF-12) Mental Scale (Norm Based)
Description: as for outcome 2
Time Frame: Baseline, Post-Intervention (3 months after baseline), Follow-Up (6 months after baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Living Well | Medical Illness Education and Support Group
Number analyzed (Participants) | 124 | 118
units on a scale
  Baseline | 41.3 (11.9) | 40.7 (11.5)
  Post-intervention: number analyzed (Participants) | 105 | 107
  Post-intervention | 44.0 (11.4) | 40.5 (11.6)
  Follow-up: number analyzed (Participants) | 106 | 104
  Follow-up | 42.7 (11.5) | 41.5 (12.2)
Statistical Analysis 1: Comparison: Living Well vs Medical Illness Education and Support Group; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.563, Mixed Models Analysis

16. Secondary Outcome: Illness Management Self-Efficacy
Description: This questionnaire is based on the items used in the original Chronic Disease Self-Management Program (CDSMP) as part of that groups extensive evaluation of the curriculum. The original CDSMP measure has been shown to have strong test-retest reliability and internal consistency as well. This subscale consists of 2 items with possible responses ranging from Never (0) to Always (5). Combined scores may range from 0-10 on this subscale, higher scores indicate greater self-efficacy.
Time Frame: Baseline, Post-Intervention (3 months after baseline), Follow-Up (6 months after baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Living Well | Medical Illness Education and Support Group
Number analyzed (Participants) | 124 | 118
units on a scale
  Baseline | 5.5 (2.1) | 5.5 (2.0)
  Post-intervention: number analyzed (Participants) | 105 | 107
  Post-intervention | 6.2 (1.9) | 5.4 (2.1)
  Follow-up: number analyzed (Participants) | 106 | 104
  Follow-up | 6.0 (2.0) | 5.4 (2.0)
Statistical Analysis 1: Comparison: Living Well vs Medical Illness Education and Support Group; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.004, Mixed Models Analysis

17. Secondary Outcome: Patient Activation Measure
Description: as for outcome 6
Time Frame: Baseline, Post-Intervention (3 months after baseline), Follow up (6 months after baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Living Well | Medical Illness Education and Support Group
Number analyzed (Participants) | 124 | 118
units on a scale
  Baseline | 60.8 (15.2) | 58.8 (14.6)
  Post-intervention: number analyzed (Participants) | 105 | 107
  Post-intervention | 64.3 (14.0) | 58.9 (14.3)
  Follow-up: number analyzed (Participants) | 106 | 104
  Follow-up | 63.4 (14.6) | 60.5 (16.1)
Statistical Analysis 1: Comparison: Living Well vs Medical Illness Education and Support Group; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.727, Mixed Models Analysis

18. Secondary Outcome: Measure of Self-Management Behaviors - General Self-Management Behaviors Subscale
Description: This questionnaire is based on the items used in the original CDSMP as part of that groups extensive evaluation of the curriculum. The original CDSMP measure has been shown to have adequate psychometric properties; the range of test-retest coefficients for the original illness management scales was .56 to .92, with internal-consistency coefficients ranging from .70 to .75. The General Self-Management Behaviors Subscale consists of 2 items with responses ranging from Never (0) to Always (5). Combined scores may range from 0-10 on this subscale, higher scores indicate greater frequency of the behavior indicating greater self-management behavior.
Time Frame: Baseline, Post-Intervention (3 months after baseline), Follow up (6 months after baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Living Well | Medical Illness Education and Support Group
Number analyzed (Participants) | 124 | 118
units on a scale
  Baseline | 2.7 (1.1) | 2.3 (1.2)
  Post-intervention: number analyzed (Participants) | 105 | 107
  Post-intervention | 2.9 (1.2) | 2.6 (1.2)
  Follow-up: number analyzed (Participants) | 106 | 104
  Follow-up | 2.9 (1.2) | 2.5 (1.2)
Statistical Analysis 1: Comparison: Living Well vs Medical Illness Education and Support Group; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.446, Mixed Models Analysis

19. Secondary Outcome: Measure of Self-Management Behaviors - Making Better Use of Health Care Subscale
Description: This questionnaire is based on the items used in the original CDSMP as part of that groups extensive evaluation of the curriculum. The original CDSMP measure has been shown to have adequate psychometric properties; the range of test-retest coefficients for the original illness management scales was .56 to .92, with internal-consistency coefficients ranging from .70 to .75. The Making Better Use of Health Care Subscale consists of 4 items with responses ranging from Never (0) to Always (5). Scores may range from 0-20 on this subscale, higher scores indicate greater frequency of behavior indicating greater self-management behavior.
Time Frame: Baseline, Post-Intervention (3 months after baseline), Follow-up (6 months after baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Living Well | Medical Illness Education and Support Group
Number analyzed (Participants) | 124 | 118
units on a scale
  Baseline | 2.9 (1.4) | 2.5 (1.4)
  Post-intervention: number analyzed (Participants) | 105 | 107
  Post-intervention | 3.3 (1.2) | 2.9 (1.3)
  Follow-up: number analyzed (Participants) | 106 | 104
  Follow-up | 3.3 (1.3) | 3.0 (1.3)
Statistical Analysis 1: Comparison: Living Well vs Medical Illness Education and Support Group; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.459, Mixed Models Analysis

20. Secondary Outcome: Measure of Self-Management Behaviors - Behavioral and Cognitive Symptom Management Subscale
Description: This questionnaire is based on the items used in the original CDSMP as part of that groups extensive evaluation of the curriculum. The original CDSMP measure has been shown to have adequate psychometric properties; the range of test-retest coefficients for the original illness management scales was .56 to .92, with internal-consistency coefficients ranging from .70 to .75. The Behavioral and Cognitive Symptom Management Subscale consists of 6 items with responses ranging from Never (0) to Always (5). Scores may range from 0-30 on this subscale, higher scores indicate greater frequency of using the behavior indicating greater self-management behavior.
Time Frame: Baseline, Post-Intervention, Follow-up (6 months after baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Living Well | Medical Illness Education and Support Group
Number analyzed (Participants) | 124 | 118
units on a scale
  Baseline | 2.2 (1.1) | 2.2 (1.0)
  Post-intervention: number analyzed (Participants) | 105 | 107
  Post-intervention | 2.5 (1.0) | 2.2 (0.9)
  Follow-up: number analyzed (Participants) | 106 | 104
  Follow-up | 2.5 (1.1) | 2.3 (0.9)
Statistical Analysis 1: Comparison: Living Well vs Medical Illness Education and Support Group; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.038, Mixed Models Analysis

21. Secondary Outcome: Measure of Self-Management Behaviors - Accessing Social Support Subscale
Description: This questionnaire is based on the items used in the original CDSMP as part of that groups extensive evaluation of the curriculum. The original CDSMP measure has been shown to have adequate psychometric properties; the range of test-retest coefficients for the original illness management scales was .56 to .92, with internal-consistency coefficients ranging from .70 to .75. The Accessing Social Support Subscale consists of 2 items with responses ranging from Never (0) to Always (5). Combined scores may range from 0-10 on this subscale, higher scores indicate greater frequency of using the behavior indicating greater self-management behavior.
Time Frame: Baseline, Post-Intervention (3 months after baseline), Follow-up (6 months after baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Living Well | Medical Illness Education and Support Group
Number analyzed (Participants) | 124 | 118
units on a scale
  Baseline | 2.3 (1.4) | 2.3 (1.2)
  Post-intervention: number analyzed (Participants) | 105 | 107
  Post-intervention | 2.4 (1.3) | 2.4 (1.3)
  Follow-up: number analyzed (Participants) | 106 | 104
  Follow-up | 2.2 (1.3) | 2.3 (1.3)
Statistical Analysis 1: Comparison: Living Well vs Medical Illness Education and Support Group; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.238, Mixed Models Analysis

22. Secondary Outcome: Measure of Self-Management Behaviors - Physical Activity Subscale
Description: This questionnaire is based on the items used in the original CDSMP as part of that groups extensive evaluation of the curriculum. The original CDSMP measure has been shown to have adequate psychometric properties; the range of test-retest coefficients for the original illness management scales was .56 to .92, with internal-consistency coefficients ranging from .70 to .75. The Physical Activity Subscale consists of 2 items with responses ranging from Never (0) to Always (5). Combined scores may range from 0-10 on this subscale, higher scores indicate greater frequency of using the behavior indicating greater self-management.
Time Frame: Baseline, Post-Intervention (3 months after baseline), Follow-up (6 months after baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Living Well | Medical Illness Education and Support Group
Number analyzed (Participants) | 124 | 118
units on a scale
  Baseline | 2.3 (1.3) | 2.3 (1.3)
  Post-intervention: number analyzed (Participants) | 105 | 107
  Post-intervention | 2.7 (1.3) | 2.4 (1.3)
  Follow-up: number analyzed (Participants) | 106 | 104
  Follow-up | 2.8 (1.3) | 2.2 (1.3)
Statistical Analysis 1: Comparison: Living Well vs Medical Illness Education and Support Group; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.011, Mixed Models Analysis

23. Secondary Outcome: Measure of Self-Management Behaviors - Healthy Eating Subscale
Description: This questionnaire is based on the items used in the original CDSMP as part of that groups extensive evaluation of the curriculum. The original CDSMP measure has been shown to have adequate psychometric properties; the range of test-retest coefficients for the original illness management scales was .56 to .92, with internal-consistency coefficients ranging from .70 to .75. The Healthy Eating Subscale consists of 2 items with responses ranging from Never (0) to Always (5).Combined scores may range from 0-10 on this subscale, higher scores indicate greater frequency of using the behavior indicating greater self-management behavior.
Time Frame: Baseline, Post-Intervention (3 months after baseline), Follow-up (6 months after baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Living Well | Medical Illness Education and Support Group
Number analyzed (Participants) | 124 | 118
units on a scale
  Baseline | 2.6 (1.3) | 2.5 (1.3)
  Post-intervention: number analyzed (Participants) | 105 | 107
  Post-intervention | 3.0 (1.1) | 2.7 (1.1)
  Follow-up: number analyzed (Participants) | 106 | 104
  Follow-up | 2.9 (1.1) | 2.8 (1.2)
Statistical Analysis 1: Comparison: Living Well vs Medical Illness Education and Support Group; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.709, Mixed Models Analysis

24. Other Pre Specified Outcome: Morisky Medication Adherence Scale
Description: This 4 item self-reported medication adherence scale was developed from a well validated 8-item scale with responses ranging from Never (0) to Very Often (4) to to better capture barriers surrounding adherence behavior. This new scale has demonstrated psychometric properties. Possible scores range from 0 to 16, with higher scores indicating greater adherence. The distribution was skewed so a square root transformation was applied before analysis.
Time Frame: Baseline, Post-intervention (3 months after baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Living Well | Medical Illness Education and Support Group
Number analyzed (Participants) | 124 | 118
units on a scale
  Baseline | 1.4 (1.0) | 1.5 (0.8)
  Post-intervention: number analyzed (Participants) | 105 | 107
  Post-intervention | 1.2 (1.0) | 1.5 (0.9)
Statistical Analysis 1: Comparison: Living Well vs Medical Illness Education and Support Group; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.134, Mixed Models Analysis

25. Other Pre Specified Outcome: Multidimensional Health Locus of Control (HLOC)
Description: Measured with a subscale of the Multidimensional Health Locus of Control. Possible scores range from 0 to 36, with higher scores indicating greater internal locus of control. An 18 item questionnaire with responses ranging on a 6 point Likert scale from Strongly Disagree to Strongly Agree that asks about self-perceived control over one's health, illnesses, and ability to take an active role in one's health.
Time Frame: Baseline, Post-intervention (3 months after baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Living Well | Medical Illness Education and Support Group
Number analyzed (Participants) | 124 | 118
units on a scale
  Baseline | 26.4 (5.9) | 26.1 (5.9)
  Post-intervention: number analyzed (Participants) | 105 | 107
  Post-intervention | 27.0 (4.8) | 25.5 (6.3)
Statistical Analysis 1: Comparison: Living Well vs Medical Illness Education and Support Group; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.045, Mixed Models Analysis

26. Other Pre Specified Outcome: Maryland Assessment of Recovery Scale (MARS)
Description: The MARS a 25-item self-report measure of recovery. Items are rated on a 5-point Likert scale ranging from not at all (1) to very much (5). The MARS has been shown to have good internal consistency (alpha=.95) and test-retest reliability (r = .868). Combined scores may range from 25-125, higher scores indicate greater self-reported recovery.
Time Frame: Baseline, Post-intervention (3 months after baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Living Well | Medical Illness Education and Support Group
Number analyzed (Participants) | 124 | 118
units on a scale
  Baseline | 3.9 (0.7) | 3.8 (0.7)
  Post-intervention: number analyzed (Participants) | 105 | 107
  Post-intervention | 4.0 (0.7) | 3.8 (0.7)
Statistical Analysis 1: Comparison: Living Well vs Medical Illness Education and Support Group; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.099, Mixed Models Analysis

27. Other Pre Specified Outcome: Morisky Medication Adherence Scale
Description: Possible scores range from 0 to 16, with higher scores indicating greater adherence. The distribution was skewed so a square root transformation was applied before analysis.
Time Frame: Baseline, Follow-up (6 months after baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Living Well | Medical Illness Education and Support Group
Number analyzed (Participants) | 124 | 118
units on a scale
  Baseline | 1.4 (1.0) | 1.5 (0.8)
  Post-intervention: number analyzed (Participants) | 105 | 107
  Post-intervention | 1.2 (1.0) | 1.5 (0.9)
  Follow-up: number analyzed (Participants) | 106 | 104
  Follow-up | 1.2 (1.0) | 1.4 (0.9)
Statistical Analysis 1: Comparison: Living Well vs Medical Illness Education and Support Group; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.852, Mixed Models Analysis

28. Other Pre Specified Outcome: Multidimensional Health Locus of Control (HLOC)
Description: as for outcome 25
Time Frame: Baseline, Post-Intervention (3 months after baseline), Follow-up (6 months after baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Living Well | Medical Illness Education and Support Group
Number analyzed (Participants) | 124 | 118
units on a scale
  Baseline | 26.4 (5.9) | 26.1 (5.9)
  Post-intervention: number analyzed (Participants) | 105 | 107
  Post-intervention | 27.0 (4.8) | 25.5 (6.3)
  Follow-up: number analyzed (Participants) | 106 | 104
  Follow-up | 26.6 (5.4) | 25.7 (5.5)
Statistical Analysis 1: Comparison: Living Well vs Medical Illness Education and Support Group; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.285, Mixed Models Analysis

29. Other Pre Specified Outcome: Maryland Assessment of Recovery Scale (MARS)
Description: The MARS a 25-item self-report measure of recovery. Items are rated on a 5-point Likert scale of not at all (1) to very much (5). Combined scores may range from 25-125, higher scores indicate greater self-reported recovery. The MARS has been shown to have good internal consistency (alpha=.95) and test-retest reliability (r = .868)
Time Frame: Baseline, Post-Invention (3 months after baseline), Follow-up (6 months after baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Living Well: Living Well (LW) will be implemented as a 12-session, peer-led, group intervention (4-8 persons) designed to help veterans with co-occurring Serious Mental Illnesses and Chronic Medical Conditions learn techniques for better health management and ways to live a healthier lifestyle. Key topics that will be discussed are medication side effects, how symptoms of mental illness may affect veterans' ability to manage their medical conditions, effects of substance use on medical and mental health functioning, learning ways to eat healthier, and how to communicate more effectively with care providers. Groups will meet weekly for 75 minutes for three months (12 sessions). There will be 3 booster sessions after the 12 sessions, once a month for 3 months.
Arm/Group | Living Well | Medical Illness Education and Support Group
Number analyzed (Participants) | 124 | 118
units on a scale
  Baseline | 3.9 (0.7) | 3.8 (0.7)
  Post-intervention: number analyzed (Participants) | 105 | 107
  Post-intervention | 4.0 (0.7) | 3.8 (0.7)
  Follow-up: number analyzed (Participants) | 106 | 104
  Follow-up | 4.0 (0.7) | 3.8 (0.7)
Statistical Analysis 1: Comparison: Living Well vs Medical Illness Education and Support Group; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.222, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Adverse events assessed from time of enrollment to follow-up assessment (~9 months) for each participant. Total duration of reported events during recruitment and follow-up of study assessments is about 2 years, 8 months.
Description: The reported All-Cause Mortality Affected and At Risk is zero as this study was deemed minimal risk and mortality due to study participation was not anticipated. In addition, there were no unanticipated deaths due to study participation.
Arm/Group | Living Well | Medical Illness Education and Support Group
All-Cause Mortality (participants affected / at risk) | 0/124 | 0/118
Serious Adverse Events (participants affected / at risk) | 0/124 | 0/118
Other Adverse Events (participants affected / at risk) | 39/124 | 30/118
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Living Well (N=124) | Medical Illness Education and Support Group (N=118)
Hospitalization (General disorders) | 39 (53) | 30 (39) — Medical or mental health hospitalizations reported during assessment, over the phone, or in group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2015-05-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT01676909/Prot_000.pdf